CLINICAL TRIAL: NCT03153605
Title: The Correlation and Relationship Between Chromaticity Parameters and Treatment Satisfaction Before and After Tooth Bleaching
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Fujian Medical University (Other)
Responsible Party: Principal Investigator, Hao Yu, Deputy Director, Department of Scientific Research, Fujian Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 201502311
Record Dates: First submitted 2017-04-24; First posted 2017-05-15 (Actual); Last update posted 2017-09-29 (Actual); Status verified 2017-05

CONDITIONS: Bleaching; Satisfactory

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SATISI_7 (Experimental)
  Interventions: Other: Common toothpaste

INTERVENTIONS:
Other: Common toothpaste — different toothpaste

SUMMARY:
Explore the correlation and specific relationship between chromaticity parameters and treatment satisfaction before and after tooth bleaching, compare the curative effect of different tooth bleaching programs.

ELIGIBILITY:
Inclusion Criteria:

* age around 20~28 years,
* at least six anterior teeth without restorations,
* good general and oral health (no dental caries and periodontal disease).

Exclusion Criteria:

* tooth sensitivity,
* any condition that could cause tooth sensitivity (non-carious cervical lesions, dentin exposure),
* participants under orthodontic treatment,
* smokers.

Ages: 20 Years to 28 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2017-10-09 (Estimated); Study Completion 2017-12-09 (Estimated)

PRIMARY OUTCOMES:
Changes of tooth color | baseline, 7 days after treatment, 14 days after treatment
  The certain points of tooth color

IPD SHARING:
Plan to Share IPD: Undecided